CLINICAL TRIAL: NCT06831591
Title: Dubousset Functional Test: An Investigation of Its Validity and Reliability in Children With GMFCS I-II Spastic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Betul Ergun, research assistant, Inonu University
Other Study IDs: Dobousset
Record Dates: First submitted 2025-02-06; First posted 2025-02-18 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy (CP); Reliability and Validity; Functional Test; Gross Motor Function Classification System (GMFCS) Level I,II
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- gmfcs 1-2: It was conducted on individuals diagnosed with spastic CP at GMFCS level I-II.

SUMMARY:
the investigators hypothesize that over time, it may lead to loss of functional capacity in children with CP. In this context, our study aims to examine the validity and reliability of the four-component Dubousset Functional Test (DFT), which is used to objectively measure the functional capacity of children with spastic CP, in children with spastic cerebral palsy at Gross Motor Function Classification System (GMFCS) I-II level.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a group of permanent disorders in the development of movement and posture due to damage to the fetal or infant brain that is not progressive but leads to limitations in activity and participation over time (Rosenbaum et al, 2007). Although the lesion in CP is not progressive, children's participation in daily life activities and social roles is limited due to secondary problems. In this sense, CP is the childhood problem that occurs in childhood and limits mobility the most (McIntyre et al, 2022).

According to the most recent classification, CP is divided into four categories: spastic, ataxic, dyskinetic and unclassifiable (Cans, C. (2000). Although spastic type CP is characterized with spasticity and hypertonus, various disorders such as weakness in muscle strength, selective motor loss, bilateral coordination failure, sensory problems, mirror movements, and inadequacy in trunk control may be observed (Cans et al., 2007). Hemiplegic spastic CP is a type in which the right or left half of the body is affected and the upper extremities are affected more than the lower extremities (Kitai et al, 2016 ). It is reported that there are 18 million children with CP worldwide and 200 thousand children with CP in Turkey and approximately 75%-85% of them have spastic CP (Cerebral Palsy Guide, 2024). In this sense, spastic CP is the most common type.

In children with spastic CP, spasticity is generally observed in the muscles of the extremities and hypotonia is generally observed in the trunk muscles. The muscles in which spasticity is most commonly observed include shoulder extensor, shoulder adductor and shoulder internal rotator muscles, elbow flexor muscles, forearm pronator muscles, wrist and finger flexor muscles, hip flexor, adductor and internal rotator muscles, knee flexor muscles and ankle plantar flexor muscles (Davids et al.).

In children with spastic CP, co-contraction of antagonist and agonist muscles is preserved instead of normal reciprocal relaxation (Aloraini et al, 2020). Although spasticity is the prominent feature, many problems such as stereotypic movement patterns, increased deep tendon reflexes, hyperreflexia and clonus, inadequacy in balance and protective reactions, combined reactions, selective motor control impairment, and decreased active and passive normal range of motion are associated. Increased muscle tone also causes secondary joint deformities, muscle contractures, posture and gait disorders. The most common types in children with spastic CP are as follows; 30-40% diparetic, 20-30% hemiparetic and 10-15% quadriparetic type CP (Vova, J. 2022).

1. Dubousset Functional Test (DFT): A conceptual four-component global functional assessment test - Dubousset Functional Test (DFT) - will be applied to objectively measure the functional capacity of children with spastic cerebral palsy (Diebo et al, 2019). These four components are as follows.

1. Get Up and Walk Test: Children with spastic cerebral palsy will get up unassisted from a seated position in a chair without arms, walk 5 meters (500 cm), turn around, walk back 5 meters and sit down again unassisted.
2. Step Test: Children with spastic cerebral palsy will climb three steps of stairs from a starting position 50 cm away, turn around on the third step and walk back down.
3. Sit and stand test: Children with spastic cerebral palsy will sit on the floor from a standing position with assistance if necessary and stand up again with assistance if necessary.
4. Dual Task Test: Children with spastic cerebral palsy will walk 5 meters forward, turn around and walk 5 meters backward while doing a memory exercise (counting down from 50 in 2 intervals).

Patients will rest for 1 hour and Dubousset Functional Test will be performed again.

2. Gross Motor Function Classification System (GMFCS) Gross motor function classification system. Developed in 1997 by Palisano et al. It was found to be valid and reliable in individuals with cerebral palsy (Palisano, 1997). Günel et al. translated the Turkish version and the evaluation form is available on the online website (Palisano, 2007).

The GMFCS used for CP is based on the child's self-initiated movement, focusing on sitting, shifting and mobility. In the five-level system, the significance of the observed differences in daily life is the main criterion. Differences are based on functional limitations, the need for hand-held mobility aids (walker, crutches or cane) or a wheelchair, and partly on the quality of movement. Expanded in 2007, the GMFCS covers the age range 12-18 years and emphasizes the World Health Organization (WHO) international classification concepts of function, disability and health (Palisano, 2007).

General characteristics of the levels

* LEVEL-1: Can walk without limitation.
* LEVEL-2: Experiences some limitations while walking.
* LEVEL-3: Walks with hand-held mobility aids.
* LEVEL-4: Movement alone is limited; may need a motorized mobility device.
* LEVEL-5: Moves with assistance in a manual wheelchair.

Statistical Method IBM SPSS 24.0 (Mac version) will be used for statistical analysis. Mean and standard deviation will be used for descriptive quantitative data and numbers and percentages will be used for qualitative data. The suitability of the data for normal distribution will be determined by Kolmogrov-Smirnov test. Repeated Measurements ANOVA, One Way ANOVA and Tukey HSD tests will be used for multiple comparisons. Chi-square test will be used in the statistical evaluation of categorical variables (frequency, percentage calculation). Significance level will be accepted as p<0.05.

The test-retest reliability of the subcomponents of the Dubousset function test will be tested with the 2-way random effect intraclass correlation coefficient (ICC) at 95% confidence interval. The ICC results will be expressed as suggested by Bland and Altman (≤0.20 poor, 0.21-0.40 fair, 0.41-0.60 moderate, 0.61-0.80 good, and 0.81-1.00 excellent). To determine the standard error of measurement (SEM) levels and the precision of the measurements, the SEM value will be calculated using the formula SEM = SD x.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years old,
* Diagnosed with spastic cerebral palsy,
* GMFCS level I-II,
* At the appropriate cognitive level to adapt to the tests to be performed in the study,
* Completed primary school level,
* Individuals who agree to participate in the study will be recruited.

Exclusion Criteria:

* Bone and/or soft tissue surgery on the lower extremities within the last 1 year,
* Inability to perform a task due to sensory, cognitive or other problems,
* Ataxic CP, Dyskinetic CP, Hypotonic CP, Mixed type CP groups will not be included in the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: G-Power 3.1.9.2 program was used to estimate the required sample size and it was observed that the effect obtained in the reference study was at a strong level (d = 0.731) (Lexell JE, Downham DY, 2005). As a result of the power analysis performed with the assumption that this effect size could be obtained again, it was calculated that 95% statistical power would be obtained at 95% confidence level if at least 33 people were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Dubousset Functional Test | 1 days
  Investigation of the Validity and Reliability of the Dubousset Functional Test in Children with GMFCS I-II Spastic Cerebral Palsy. It is a test used to objectively measure the functional capacity of children with spastic CP. The DFT includes 4 different test components. After the patients are administered the DFT, they will rest for 1 hour and then the DFT will be administered again. The time to complete the tests will be recorded in seconds and evaluated before and after.

SECONDARY OUTCOMES:
TUG (Timed Up and Go) Test | Day 1
  The TUG test is a tool designed to assess dynamic balance, walking speed and mobility. To complete the test, participants are required to get up from a chair with armrests, walk 3 m, turn, walk back and sit on the chair. The completion time of the test is recorded with a stopwatch
Dual Task TUG (Additional Cognitive Task) | Day 1
  During the TUG test, counting backwards by twos from 50 will be used as an additional cognitive task. When the test had to be repeated, individuals continued counting from the number they had left off. Counting errors will be ignored.
Three-Meter Backward Walk Test (3MBWT) | day 1
  Participant walks backward along a 3-meter line marked with tape as quickly as possible, keeping heels aligned with the line. Completion time is measured.
Functional Reach Test | day 1
  Standing with one arm flexed to 90°, participant reaches forward as far as possible without moving the feet. The distance between the starting and farthest fingertip positions is recorded. The test is repeated three times, and the average is used.
Pediatric Balance Scale | day 1
  Balance performance is assessed using the Pediatric Balance Scale, which consists of 14 items scored from 0 to 4. Higher scores indicate better balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Physical Medicine and Rehabilitation Clinic, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ergun B, Baykan M, Baykan Copuroglu O, Abakay H, Guc A, Karabulut R. Functional motor performance and reliability of the Dubousset Functional Test in ambulatory children with spastic cerebral palsy. Dev Neurorehabil. 2026 Feb 7:1-7. doi: 10.1080/17518423.2026.2626754. Online ahead of print. PMID 41653057